CLINICAL TRIAL: NCT03672084
Title: Allogeneic Hematopoietic Stem Cell Transplantation Following Conventional Chemotherapy in High Risk Peripheral T Cell Lymphoma
Brief Title: Allo-HSCT as First-line Consolidation in High-risk PTCL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, PI, Peking University People's Hospital
Other Study IDs: Allo-HSCT for PTCL
Record Dates: First submitted 2018-09-13; First posted 2018-09-14 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Results of conventional therapy in patients with peripheral T-cell lymphoma(PTCL) are poor. Allogeneic hematopoietic stem cell transplantation(allo-HSCT) gave excellent results in PTCL after failure of conventional therapy and in many cases also of HDT/ASCT. A disadvantage of allo-HSCT is high TRM rate, especially in refractory or relapsed patients. Another limitation to the use of allo-HSCT is the availability of a HLA matched donors. Haploidentical family donors have been successfully used in treatments of hematologic malignancies, including malignant lymphomas. Thus, allo-HSCT could be used as first-line consolidation following conventional chemotherapy in high-risk PTCL patients. The study hypothesis: Using allo-HSCT as consolidation following chemotherapy in high-risk PTCL exerts a strong anti-lymphoma effect and could increase response rate and improve long term survival.

DETAILED DESCRIPTION:
After primary diagnosis eligible patients receive 2 to 3 courses of CHOEP-21 with formal restaging after course 2. Patients with CR, PR or no change proceed to allo-HSCT. Donor selection: Matched sibling donor(MSD) is the first choice. An unrelated donor or haploidentical family donor search is performed in patients without sibling donor. The primary end point was 1 year progression-free survival. The secondary end points were complete commission rate, transplant-related mortality, overall survival, relapse rate and graft-versus-host disease (GVHD) . Following time is 2 years

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of mature T-cell lymphoma, stage 2-4, or stage 1 with aa IPI>=0
* age <= 60 years
* KPS>=70

Exclusion Criteria:

* stage I with aaIPI 0, ALCL ALK positive, T-lymphoblastic lymphoma, cutaneous T-cell lymphoma
* HIV positivity
* major organ dysfunction
* pregnancy
* patient unable to give informed consent

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Mature T-cell lymphoma patietnts, stage 2-4, or stage 1 with aa IPI>=0
  * age <= 60 years
  * KPS>=70
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
1 year PFS | participants will be follow for an expected average of 365 days
  progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Jun Huang, MD, Principal Investigator — Peking University
Locations (1):
- Peking University People's Hospital, Beijing, China